CLINICAL TRIAL: NCT00056966
Title: Phase I/II Study of CD45 Antibodies and Alemtuzumab Conditioning Regimen for Allogeneic Hematopoietic Stem Cell Transplantation of Patients With Hematological Diseases
Brief Title: Conditioning Regimen for Allogeneic Hematopoietic Stem Cell Transplantation of Patients With Hematological Diseases
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, George Carrum, Associate Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12472; ACHE; NCT00602888 (obsolete NCT alias)
Record Dates: First submitted 2003-03-26; First posted 2003-03-27 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-06

CONDITIONS: Hematologic Malignancy
Keywords: Acute myeloid leukemia; Acute lymphoblastic leukemia; Chronic myeloid leukemia; Non-Hodgkin's lymphoma; Hodgkin's disease; Myelodysplastic syndrome; Myeloproliferative disorders; Multiple myeloma; Severe aplastic anemia
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphoma, Non-Hodgkin; Hodgkin Disease; Myelodysplastic Syndromes; Myeloproliferative Disorders; Multiple Myeloma; Anemia, Aplastic | interventions — Alemtuzumab; Tacrolimus; fludarabine; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): recipients of HLA matched sibling transplants
  Interventions: Drug: ANTI-CD45; Drug: CAMPATH-1H; Drug: FK506; Drug: Fludarabine; Radiation: Total Body Irradiation; Procedure: Stem cell infusion
- 2 (Experimental): recipients of unrelated or mismatched family donor transplants
  Interventions: Drug: ANTI-CD45; Drug: CAMPATH-1H; Drug: FK506; Drug: Fludarabine; Radiation: Total Body Irradiation; Procedure: Stem cell infusion

INTERVENTIONS:
Drug: ANTI-CD45 — 400ug/kg Day-5 through Day-2
Drug: CAMPATH-1H — Day -8 through Day -6 Dosed per Institutional SOP
  Other Names: anti-CD52; alemtuzumab
Drug: FK506 — Day -2 through Day 30 dose adjusted to maintain level between 5-15 ng/ml.
  Other Names: tacrolimus
Drug: Fludarabine — Day-8 through Day-5 30 mg/m2
Radiation: Total Body Irradiation — Day-1 single dose 450 cGy
Procedure: Stem cell infusion — Patients will receive peripheral blood stem cells from a HLA matched or one antigen mismatched related or unrelated donor (target CD34+ cell count >2 x 106/kg). When peripheral stem cells are unavailable or insufficient, bone marrow (target mononuclear cell count >2 x 108/kg) will be substituted.

SUMMARY:
Participants in this study have a hematologic malignancy (a disorder in the bone marrow that affects the body's ability to create blood) that might benefit from receiving an allogeneic stem cell transplant (meaning the cells come from a donor) from a family member or nearly identical matched donor. The donor may either be a matched sibling, a mismatched family member, or an unrelated person.

Usually these patients are given high doses of chemotherapy before receiving a stem cell transplant to keep their immune system from rejecting the donor stem cells and to kill any diseased cells that remain in the body. However, this group of patients have a high risk of developing possibly life-threatening treatment-related side effects such as infections, damage to vital organs such as lungs, liver, kidney and heart, as well as graft versus host disease (GVHD).

Instead of the high dose chemotherapy and radiotherapy usually given before a transplant, this research study uses a new pre-transplant combination of three drugs, Fludarabine, Anti-CD45 and CAMPATH-1H with low dose radiotherapy. Fludarabine is a chemotherapy drug while Anti-CD45 and CAMPATH-1H are antibodies against certain types of blood cells, including those which are causing this disease. CAMPATH-1H is particularly important because it stays active in the body for a long time after it is given, which means it may work longer to prevent GVHD symptoms. Anti-CD45 may help in eradicating residual malignant cells. All these agents also help in preventing rejection of donor stem cells. This study is designed to give a less intense chemotherapy and radiotherapy, so that the life-threatening toxicities of conventional high dose chemotherapy and radiotherapy regimen can be reduced, while maintaining the ability to cure cancer.

DETAILED DESCRIPTION:
CAMPATH-1H will be given as a daily IV infusion for three days. Fludarabine will be given as a daily IV infusion for four days. Anti-CD45 will be given as a daily IV infusion for 4 days. Patients will then receive radiotherapy (also known as Total Body Irradiation or TBI) for one day. A summary of the treatment follows:

* Day - 8: CAMPATH-1H and Fludarabine
* Day - 7: CAMPATH-1H and Fludarabine
* Day - 6: CAMPATH-1H and Fludarabine
* Day - 5: Anti-CD45 and Fludarabine
* Day - 4: Anti-CD45
* Day - 3: Anti-CD45
* Day - 2: Anti-CD45
* Day - 1: TBI
* Day 0: Stem Cell Infusion (transplant)

To help prevent the body from developing GVHD, patients will also receive the drug FK506, starting two days before the transplant and continuing for at least one month.

Both the CAMPATH-1H and the Anti-CD45 can cause allergic reactions so patients will be given drugs to help prevent those reactions before receiving daily doses.

To see how CAMPATH-1H works in patients with hematologic malignancies, some patients will be asked to participate in pharmacokinetic studies. For this, approximately 13 blood samples will be taken from the central line scheduled before each infusion on Day -8 to Day -6, daily thereafter until Day 0, and then approximately once per week on days 7, 14, 21 and 28 post transplant. No more than 5 teaspoonfuls total will be drawn.

To see how Anti-CD45 works in patients with hematologic malignancies some patients will be asked to participate in pharmacokinetic studies. Approximately 22 blood samples will be taken from the central line scheduled before, during and after each infusion and after the end of the last infusion of Anti-CD45. No more than 10 teaspoonfuls total will be drawn over the course of the four anti-CD45 infusions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with one of the following high risk diseases needing allogeneic hemopoietic stem cell transplantation:

   Acute myeloid leukemia either a) Primary refractory, or b) Beyond first complete remission(CR1), or c) In CR1 with high risk of relapse

   Acute lymphoblastic leukemia either a) Primary refractory, or b) Beyond first complete remission(CR1), or c) In CR1 with high risk of relapse

   Chronic myeloid leukemia, either a) Accelerated phase, or b) Blast crisis, or c) Chronic phase and not achieving major cytogenetic response despite standard therapy

   Chronic lymphocytic leukemia, either a) Primary refractory, or b) Beyond first complete remission(CR1),

   Non Hodgkin's lymphoma, either a) Primary refractory, or b) Beyond first complete remission(CR1)

   Hodgkin's disease, either a) Primary refractory, or b) Beyond first complete remission(CR1),

   Myelodysplastic syndrome with IPSS score > 0. (Appendix A)

   Myeloproliferative disorders (with the exclusion of chronic myeloid leukemia) a) Primary Myelofibrosis with Lile score of 1 or 2 (Appendix B) b) Polycythemia Vera or Essential Thrombocythemia transformed to AML or Myelofibrosis and PV "spent phase"

   Multiple Myeloma with stage II or III disease

   Severe aplastic anemia
2. Conditions that increase Treatment Related Mortality (need one or more to be eligible):

   Greater or equal to 35 years of age;

   Ejection Fraction of less than 50%;

   DLCO less than 50% or FEV1/FVC < 80% of predicted value;

   Diabetes Mellitus;

   Renal insufficiency (serum creatinine abnormal);

   Hepatic dysfunction-transaminases, or alkaline phosphatase, or bilirubin twice the upper limit of normal;

   Prior recent history of systemic fungal infection;

   Multiple prior treatment regimens (equal to or more than 3);

   Significant Grade III or IV neurologic, cardiac, pulmonary, renal or hepatic toxicity from previous treatment;

   Prior Autologous or Allogeneic Stem Cell transplantation;
3. Available Healthy Donor without any contraindications for donation. 5/6 or 6/6 related or unrelated donor (molecular typing for DRB1);
4. Patient and/or responsible person able to understand and sign consent

Exclusion Criteria:

Pregnant and lactating women, or women unwilling to use contraception.

HIV positive patient

Unstable angina and uncompensated congestive heart failure (Zubrod of 3 or greater)

Severe chronic pulmonary disease requiring oxygen (Zubrod of 3 or greater)

Child's class C cirrhosis

Unstable cerebral vascular disease or recent hemorrhagic stroke (less than 6 months)

Patients with known allergy to rat serum products

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2002-11; Primary Completion 2005-05 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Assess safety and feasibility of monoclonal abs directed to CD45 and CD52 antigens, Fludarabine and low dose TBI, as a non-myeloablative preparatory regimen for allo HSCT. This will be determined by 100d Non-relapse mortality and 100d Graft rejection | 100 days post transplant

SECONDARY OUTCOMES:
To obtain a preliminary estimate of the efficacy of this therapy as defined by: Complete remission at day 100 and One-year disease free survival. | 100 days and 1 year post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm K Brenner, MD, Study Chair — Baylor College of Medicine
Locations (2):
- United States (2):
  - Texas Children's Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas